CLINICAL TRIAL: NCT02924636
Title: Electronic-personalized Program for Obesity in Pregnancy to Improve Delivery - ePPOP Study
Brief Title: Electronic-personalized Program for Obesity in Pregnancy to Improve Delivery
Acronym: ePPOP-ID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2015_03; 2015-A00937-42 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2016-10-04; First posted 2016-10-05 (Estimated); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Obesity; Pregnancy
Keywords: C-section; Instrumental delivery; Pregnancy complications; Macrosomia; Neonatal complications
MeSH Terms: conditions — Obesity; Pregnancy Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): personalized and online intervention. The intervention website will provide secure communication with dietician and lifestyle coaches. Women will receive emails and monthly newsletters with new content and reminder.
  Interventions: Behavioral: ePPOP-ID program
- Control (No Intervention): standard care with oral information about the goal of nutritional needs during pregnancy and gestational weight gain guidelines according to BMI

INTERVENTIONS:
Behavioral: ePPOP-ID program — This is a personalized and online program. The website will provide secure communication with dietician and lifestyle coaches.
  Arms: Intervention

SUMMARY:
The purpose of this study is to assess the efficacy of an electronic-based intervention to help pregnant overweight and obese women gain an appropriate amount of weight and improve their delivery i.e. to reduce the rate of labour procedures and interventions. We chose a composite outcome including instrumental delivery and Caesarean section, as clinically relevant outcomes because the mode of delivery is one of the major goals of the obstetrical management and is is strongly associated with body mass index and gestational weight gain.

DETAILED DESCRIPTION:
Our study is an open, multicenter, randomized, parallel-group, controlled trial. This study will include obese pregnant women recruited in 11 French university hospitals. Patients will be randomized into two-parallel groups. One group underwent the electronic-personalized program (the interventional group) and the other underwent standard care (the control group). Due to the intervention by itself, a blind study would not be achievable.

Intervention group (the electronic-personalized program) The intervention will be presented as a comprehensive dietary and lifestyle intervention called "e-PPOP-ID" (electronic Personalized Programmed for Obesity in Pregnancy to Improve Delivery), including a combination of dietary, exercise, and behavioral strategies delivered on a web site.

The intervention will start at the latest by 20 weeks of pregnancy throughout the pregnancy and 8 weeks post-partum.

Pregnant women of the intervention group will be given an access to a personalized patient centric e-health platform. The platform we be specifically designed for this program. Various modules of this platform will be activated:

- An e-learning program: An e-Learning module will propose personalized content to each patient. Before the program, patients have to fill in questionnaires about food consumption (FFQ), Eating behavior (TFEQ) and physical activity (IPAQ). The answers of these questionnaires will be taken into account to define the e-learning lessons that patients must follow.Multi educational supports such as videos, fact sheets, quiz will be integrated into this program. Patient will be motivated to validate their program thanks to a reward system (access to new content by earning stars) and their knowledge can be estimated thanks to a quiz system.

Dieticians and adapted physical education teachers will develop the content.These lessons will include nutritional needs, motivational and behavioral advices, recipes, and movies of exercises easily achievable. The objective e-learning program is to limit weight gain by encouraging to healthy balance of carbohydrates, fat, protein, reducing high-energy foods intake (refined carbohydrates and saturated fats), increasing intake of fruits and vegetables and also by encouraging to physical activity. A second evaluation at around the 30th gestational weeks will allow adapting the lessons of the e-learning program, according to the progress of patients.

A Social network:

The platform will propose various social networking tools that can link the patient together or link the patient with the care team. Using a pseudo, patient will be able to connect together and interact with various tools such as a secured instant message system, a secured videoconference and a forum.

Motivation concepts Pregnant women will receive emails, which will encourage them to log in website and follow an e-learning lessons.A newsletter will be sent every month and will link to the new contents of the web site.Adhesion of program will be measured monthly by self-questionnaire of satisfaction and by measuring the time spent on the website including the forum.

Control group (Standard care):

The control group will receive standard care with oral information about the goal of nutritional needs during pregnancy and gestational weight gain guidelines according to BMI.

ELIGIBILITY:
Inclusion Criteria:

* Obese pregnant women (30 ≤ BMI < 40 kg/m2)
* Singleton pregnancy between 12+0 to 19+6 weeks of pregnancy
* Having an email address and an Internet access

Exclusion Criteria:

* BMI < 30 kg/m2 or BMI > 40 kg/m2
* History of more than 2 miscarriages
* Severe heart disease (arrhythmias, history of myocardial infarction)
* Multiple pregnancy
* Unstable thyroid disease
* Uncontrolled hypertension
* Pre-gestational diabetes
* Bariatric surgery
* Any medical condition that may interfere with physical activity during pregnancy
* No access to Internet
* Minor
* Absence of health insurance
* Guardianship
* Refusal to participate in research

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 857 (Actual)
Dates: Start 2017-11-13 (Actual); Primary Completion 2022-03-13 (Actual); Study Completion 2022-04-13 (Actual)

PRIMARY OUTCOMES:
rate of obstetrical interventions | at birth
  Caesarean section and instrumental delivery (forceps and vacuum extractor)

SECONDARY OUTCOMES:
Total gestational weight gain | at birth
Gestational hypertension | at birth
  blood pressure > 140 and/or 90 mmHg after 20 weeks
Preeclampsia | at birth
  gestational hypertension and proteinuria = 0.30 g/24 h
Gestational diabetes mellitus | at birth
  Diagnosed by a 75g-oral glucose tolerance test (OGTT) between 24 and 28 according to French guidelines and International Association diabetic and Pregnancy Study Group
Premature birth | at birth
gestational age | at birth
Birth weight | at birth
Apgar score | at birth
Arterial umbilical cord pH | at birth
Neonatal traumatism | at birth
  composite outcome (shoulder dystocia + fracture + brachial plexus injury)
Hyperbilirubinemia | 1st week after birth
Neonatal respiratory distress syndrome | 1st week after birth
Transfer in neonatal intensive care unit | 1st week after birth
Maternal fever | 1st week after delivery
Thromboembolic event | 1st week after delivery
Hemorrhage | 1st week after delivery
Breastfeeding duration | 8 weeks +/- 2 weeks after delivery
Maternal weight | 8 weeks +/- 2 weeks after delivery
child weight | 8 weeks +/- 2 weeks after delivery

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Deruelle, MD, PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- CHU Lille, Lille, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Deruelle P, Lelorain S, Deghilage S, Couturier E, Guilbert E, Berveiller P, Senat MV, Vayssiere C, Sentilhes L, Perrotin F, Gallot D, Chauleur C, Sananes N, Roth E, Luton D, Caputo M, Lorio E, Chatelet C, Couster J, Timbely O, Doret-Dion M, Duhamel A, Pigeyre M. Rationale and design of ePPOP-ID: a multicenter randomized controlled trial using an electronic-personalized program for obesity in pregnancy to improve delivery. BMC Pregnancy Childbirth. 2020 Oct 7;20(1):602. doi: 10.1186/s12884-020-03288-x. PMID 33028261